CLINICAL TRIAL: NCT07076277
Title: Visual Outcomes in Patients Contralaterally Implanted With PanOptix Pro and Clareon Vivity Compared to Bilateral Implantation of PanOptix Pro
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Brian Shafer (Other)
Responsible Party: Sponsor-Investigator, Brian Shafer, Ophthalmologist, Shafer Vision Institute
Organization: Shafer Vision Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SVI-POPCV-001
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cataract; Multifocal Intraocular Lens
Keywords: multifocal intraocular lens; cataract; cataract surgery; Presbyopia Correcting IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking: Double (Participant, Outcomes Assessor) Masking Description: Subjects and outcomes assessors will be blinded to IOL assignments to reduce bias in patient-reported outcomes and visual acuity testing. Surgeons are unmasked for implantation procedures but do not participate in postoperative assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Contralateral PanOptix Pro and Clareon Vivity (Experimental): Subjects randomized to this arm will receive bilateral cataract surgery with contralateral implantation: Alcon Clareon PanOptix Pro or PanOptix Pro Toric IOL in one eye and Alcon Clareon Vivity or Vivity Toric IOL in the fellow eye. The Vivity IOL will be implanted in the dominant eye, with all surgeries targeting emmetropia. Residual astigmatism will be managed to ≤0.50 diopters using toric IOLs or arcuate incisions as needed.
  Interventions: Device: Clareon PanOptix Pro and Clareon Vivity Intraocular Lens
- Bilateral PanOptix Pro (Active Comparator): Subjects randomized to this arm will receive bilateral cataract surgery with implantation of Alcon Clareon PanOptix Pro or PanOptix Pro Toric IOLs in both eyes. All eyes will be targeted for emmetropia, and residual astigmatism will be controlled to ≤0.50 diopters using toric IOLs or arcuate incisions as appropriate.
  Interventions: Device: Clareon PanOptix Pro Intraocular Lenses

INTERVENTIONS:
Device: Clareon PanOptix Pro and Clareon Vivity Intraocular Lens — Bilateral cataract surgery with contralateral implantation: Alcon Clareon PanOptix Pro (or PanOptix Pro Toric) intraocular lens in one eye and Alcon Clareon Vivity (or Vivity Toric) intraocular lens i
  Arms: Contralateral PanOptix Pro and Clareon Vivity
Device: Clareon PanOptix Pro Intraocular Lenses — Bilateral cataract surgery with implantation of Alcon Clareon PanOptix Pro (or PanOptix Pro Toric) intraocular lenses in both eyes. All surgeries target emmetropia with residual astigmatism ≤0.50 diopters using toric IOLs or arcuate incisions as needed.
  Arms: Bilateral PanOptix Pro

SUMMARY:
Title:

Visual Outcomes in Patients Contralaterally Implanted with PanOptix Pro and Clareon Vivity Compared to Bilateral Implantation of PanOptix Pro

Sponsor:

Brian Shafer, MD, Shafer Vision Institute

Objective:

To compare visual outcomes and patient-reported satisfaction in cataract patients receiving either:

Contralateral implantation (PanOptix Pro in one eye, Clareon Vivity in the other)

Bilateral PanOptix Pro implants

Key hypotheses:

Contralateral implantation is non-inferior for binocular best-corrected distance visual acuity (BCDVA) at 4 m.

Contralateral implantation yields superior visual disturbance outcomes (less halo, glare, starburst).

Design:

Prospective, randomized, double-masked, two-arm, multicenter study

N = 346 subjects (173 per arm)

5 surgeons across 4 sites

All patients undergo bilateral phacoemulsification aiming for emmetropia

Randomized 1:1 to:

Arm 1: PanOptix Pro (dominant eye) + Clareon Vivity (non-dominant eye)

Arm 2: Bilateral PanOptix Pro

Surgical Details:

Femtosecond laser optional

Second eye surgery ≤4 weeks after first

Toric IOLs or arcuate incisions for residual astigmatism ≤0.50 D

Biometry with ARGOS, IOLMaster 700, or Lenstar

Toric alignment with ORA, Callisto, etc.

Assessments:

Visual acuity at 4 m, 66 cm, 40 cm, 33 cm in photopic and mesopic conditions

Defocus curves, contrast sensitivity (with/without glare)

Manifest refraction

Patient-reported outcomes via IOLSAT and QUVID questionnaires

Masking: subjects and assessors unaware of IOL assignments

Endpoints (at 3 months):

Primary: Binocular BCDVA (4 m)

Secondary: DCIVA, DCNVA, UDVA, UIVA, UNVA, defocus curves, refractive outcomes, visual disturbance scores

Exploratory: Mesopic VA, low contrast VA, contrast sensitivity, satisfaction scores

Eligibility Criteria:

Adults with bilateral age-related cataracts

Plan for bilateral phacoemulsification

Expected postop monocular BCDVA ≤0.1 logMAR (20/25)

Residual astigmatism ≤0.50 D

Exclusions include corneal pathology, macular disease, glaucoma, prior ocular surgery, amblyopia, severe dry eye, high HOA (>0.6 um), monovision preference, active infection/inflammation, pregnancy

Statistics:

Non-inferiority margin: 0.1 logMAR

Superiority testing for visual disturbances

Step-down testing hierarchy for primary and secondary outcomes

Sample size powered for 80% at α=0.05, accounting for 10% dropout

Two-proportion Z-tests for dysphotopsia rates

Safety Monitoring:

Adverse Events (AEs) and Serious Adverse Events (SAEs) captured

Definitions, severity grading, and reporting procedures specified

Protocol deviations documented and reported per IRB requirements

Data Handling:

Data anonymized via subject numbers

Stored securely (locked cabinets, password-protected systems)

Study registered at ClinicalTrials.gov

Visit Schedule:

Screening: Consent, eligibility, history

1st & 2nd Eye Surgery Visits

3-Month Post-Op Visit: Comprehensive visual assessments, questionnaires, AE review

DETAILED DESCRIPTION:
SVI-POPCV-001 Protocol Detailed Description

Title:

Visual Outcomes in Patients Contralaterally Implanted with PanOptix Pro and Clareon Vivity Compared to Bilateral Implantation of PanOptix Pro

Sponsor and Investigator Brian Shafer, MD

Shafer Vision Institute, USA

Study Phase: Investigator-Initiated Trial (IIT)

RTI#: 25-IL73, IIT Proposal #97074289

Protocol Version 1.0 (21 May 2025)

Study Objective

To evaluate visual outcomes and patient-reported satisfaction in patients with bilateral age-related cataracts randomized to either:

Contralateral implantation (PanOptix Pro in one eye and Clareon Vivity in the other)

Bilateral PanOptix Pro implantation

Hypotheses:

Contralateral approach will be non-inferior in binocular BCDVA at 4 m.

Contralateral approach will yield superior outcomes in reducing visual disturbances like halos.

Study Design Prospective, randomized, double-masked, two-arm, multicenter trial

5 surgeons at 4 sites

N=346 subjects (173 per arm), powered for 80% with 10% dropout buffer

Randomized 1:1

Arm 1: PanOptix Pro (dominant eye) + Clareon Vivity (non-dominant eye)

Arm 2: Bilateral PanOptix Pro

All surgeries target emmetropia

Surgical Methods Bilateral phacoemulsification

Optional femtosecond laser-assisted cataract surgery

Second eye surgery within 4 weeks

Residual astigmatism ≤0.50 D, managed with toric IOLs or arcuate incisions

Preoperative IOL calculation using Barrett Universal II and Barrett Toric Calculator

Toric alignment via ORA, Veracity, or digital/femtosecond laser marking

Biometry with ARGOS, IOLMaster 700, Lenstar

HOA/coma measurement with topography (Cassini, Pentacam, iTrace, Atlas)

Assessment Tools M&S Clinical Trial Suite (CTS) for standardized VA testing

Validated questionnaires (IOLSAT, QUVID) for patient-reported outcomes

Measurements:

Photopic & mesopic VA

Defocus curves

Contrast sensitivity with/without glare

Manifest refraction

Masking:

Subjects and outcome assessors blinded to IOL assignment

Endpoints

Primary Endpoint (3 months):

Binocular best-corrected distance VA (BCDVA) at 4 m

Secondary Endpoints (3 months):

Binocular DCIVA at 66 cm

DCNVA at 40 cm and 33 cm

UDVA, UIVA, UNVA at the same distances

Defocus curves over ±3.00 D range

Refractive outcomes (sphere, cyl, MRSE)

Visual disturbance scores via QUVID

Exploratory:

Mesopic VA

Photopic low-contrast VA

Mesopic contrast sensitivity (with/without glare)

Patient satisfaction via IOLSAT

Eligibility

Inclusion:

Adults with bilateral age-related cataracts

Suitable for bilateral phacoemulsification

Post-op monocular BCDVA expected ≤0.1 logMAR (20/25)

Residual astigmatism ≤0.50 D

Normal ocular exam except cataract

Exclusion:

Corneal pathology or irregular astigmatism

Retinal disease, macular degeneration, glaucoma

Severe dry eye, nystagmus, strabismus

Zonular instability or pseudoexfoliation

Prior ocular surgery (including refractive)

Monovision preference

Amblyopia or monofixation

HOA >0.6 um

Combined procedures planned

Participation in conflicting trials

Pregnancy/breastfeeding

Statistical Analysis Non-inferiority margin: 0.1 logMAR

Step-down analysis order:

BCDVA (non-inferiority)

DCIVA (non-inferiority)

DCNVA 33 cm (superiority)

Visual disturbance rates (superiority) 5-9. Other VA measures (non-inferiority/superiority)

Alpha = 0.05

Two-proportion Z-test for visual disturbances

t-tests or Wilcoxon tests depending on distribution

Defocus curve comparisons via 2-way ANOVA

Sample Size Justification:

Powered for BCDVA difference of 0.05 logMAR with SD 0.15

Minimum ~250 needed accounting for dropout

Cap of ~70 subjects per surgeon, adjustable with approval

Adverse Event Management AEs: any abnormal ocular signs/symptoms

SAEs include death, life-threatening events, hospitalization, disability, congenital anomalies

Adverse Device Effects: linked to IOL or surgical process

Severity grading: mild, moderate, severe (not same as SAE)

Investigator assessment of relationship (not/possibly/probably/definitely related)

Immediate reporting of SAEs/ADEs to sponsor/IRB

Protocol deviations documented and reported per IRB policy

Data Handling Data de-identified with subject numbers

Source documents secured physically and digitally

Strict confidentiality per law

ClinicalTrials.gov registration

IRB oversight for amendments, AE/SAE reports, study closure

Confidentiality and Regulatory Compliance Results may be published without identifying participants

Data shared with sponsor, regulatory agencies, IRB

Conducted per protocol, GCP, and applicable laws

ELIGIBILITY:
Inclusion Criteria Adult patients (≥18 years old) able and willing to provide informed consent.

Bilateral diagnosis of age-related cataracts.

Planned bilateral cataract removal by phacoemulsification with either:

Contralateral implantation of Clareon PanOptix Pro/PanOptix Pro Toric in one eye and Clareon Vivity/Vivity Toric in the fellow eye, or

Bilateral implantation of Clareon PanOptix Pro/PanOptix Pro Toric.

Expected best monocular corrected distance visual acuity (BCDVA) of 0.1 logMAR (Snellen 20/25) or better in both eyes postoperatively, as determined by the surgeon.

Residual astigmatism expected to be ≤0.50 diopters in both eyes postoperatively (using toric IOLs or arcuate incisions as needed).

Normal ocular findings aside from cataracts.

Exclusion Criteria Corneal pathology or irregular astigmatism.

Preexisting macular disease or other retinal degenerative disease expected to cause vision loss.

Glaucoma.

Severe dry eye disease.

Nystagmus or strabismus.

Zonular laxity or dehiscence, pseudoexfoliation.

Any condition (in the investigator's opinion) that may affect study endpoints.

Previous history of any ocular surgery, including corneal refractive surgery.

Subjects desiring monovision.

History of amblyopia or monofixation syndrome with poor stereoscopic vision.

Total corneal higher-order aberrations (HOA) greater than 0.6 microns.

Any planned simultaneous or combined procedures at the time of cataract surgery (e.g., MIGS).

Participation in another clinical study that could interfere with study results.

Any active ocular infection or inflammation.

Pregnant, breastfeeding, or planning to become pregnant during the study (as determined by verbal inquiry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Binocular Best-Corrected Distance Visual Acuity (BCDVA) at 4 meters | 3 months post-operative visit
  Binocular BCDVA measured in logMAR under photopic conditions (85 cd/m²) at 4 m using standardized ETDRS charts with the M&S Clinical Trial Suite (CTS). Non-inferiority margin of 0.1 logMAR between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shafer, MD, Principal Investigator — Shafer Vision Institute
Locations (5):
- United States (5):
  - VIP Eye Care, Baltimore, Maryland
  - Vance Thompson Vision, Alexandria, Minnesota
  - Vance Thompson Vision, Bozeman, Montana
  - Main Line Surgery Center, Bala-Cynwyd, Pennsylvania
  - Shafer Vision Institute, Plymouth Meeting, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Not applicable; individual participant-level data will not be shared.

REFERENCES:
- [Background] Hovanesian JA, Jones M, Allen Q. The Vivity Extended Range of Vision IOL vs the PanOptix Trifocal, ReStor 2.5 Active Focus and ReStor 3.0 Multifocal Lenses: A Comparison of Patient Satisfaction, Visual Disturbances, and Spectacle Independence. Clin Ophthalmol. 2022 Jan 18;16:145-152. doi: 10.2147/OPTH.S347382. eCollection 2022. PMID 35082481
- [Background] Arrigo A, Gambaro G, Fasce F, Aragona E, Figini I, Bandello F. Extended depth-of-focus (EDOF) AcrySof(R) IQ Vivity(R) intraocular lens implant: a real-life experience. Graefes Arch Clin Exp Ophthalmol. 2021 Sep;259(9):2717-2722. doi: 10.1007/s00417-021-05245-6. Epub 2021 May 29. PMID 34050809
- [Background] Sudhir RR, Dey A, Bhattacharrya S, Bahulayan A. AcrySof IQ PanOptix Intraocular Lens Versus Extended Depth of Focus Intraocular Lens and Trifocal Intraocular Lens: A Clinical Overview. Asia Pac J Ophthalmol (Phila). 2019 Jul-Aug;8(4):335-349. doi: 10.1097/APO.0000000000000253. PMID 31403494